CLINICAL TRIAL: NCT04591340
Title: Effect of Standardized Nutrient Management on Clinical Outcomes of Hematopoientic Stem Cell Transportation Patients--a Cross-sectional Study
Brief Title: Effect of Standardized Nutrient Management on Clinical Outcomes of Hematopoientic Stem Cell Transportation Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: YYK-2020003
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Nutrition Related Cancer
Keywords: HSCT; Nutrtion
MeSH Terms: interventions — Nutrition Assessment; Dietary Supplements; Parenteral Nutrition, Total

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- test group: all the patients treated with HSCT are with nutrition risk, so they will be all included to accept nutrition therapy.
  Interventions: Dietary Supplement: dietary advice, oral nutritional supplement, supplementary parenteral nutrition or total parenteral nutrition

INTERVENTIONS:
Dietary Supplement: dietary advice, oral nutritional supplement, supplementary parenteral nutrition or total parenteral nutrition — All HSCT(hematopoietic stem cell transplantation) patients should be accepted dietary advice or oral nutritional supplement, if their energy intake will not reach 60% of the goal level during the transplanting, then supplementary parenteral nutrition or total parenteral nutrition.

SUMMARY:
To analysis a standardized stepped nutritional treatment process for patients with hematopoietic stem cell transportation, including nutritional risk screening and assessment, standardized nutritional treatment implementation, therapeutic effect follow-up and monitoring, family nutritional treatment follow-up, etc

DETAILED DESCRIPTION:
Standardized nutrition therapy for patients with hematopoietic stem cell transportation should follow the principle of sequential treatment of nutrition, which is the preferred scheme with individualized dietary advice or oral nutritional supplement, if their energy intake will not reach 60% of the goal level during the transplanting, then supplementary parenteral nutrition or total parenteral nutrition is needed. The standardized nutrition therapy aims to improve quality of life and long-term survival rate of patients, reduce the complications and social burden of disease.

ELIGIBILITY:
Inclusion Criteria:

* • Patients treated with HSCT

Exclusion Criteria:

* nothing

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Both female and male patients and between 10 to 79 years old treated with HSCT can be included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of nutritional status | 4 months
  We collect the body composition and grip strength of every HSCTpatients. Body composition include the muscle and fat contents.They are all measured as kilogram. (kg). Specific nutritional guidelines will be provided based on body composition results
Improvement of quality of life | 4 months
  We asked each patient to complete the quality of life scale for every HSCTpatient. There are 32 questions in the scale, and each question has 4-7 options. The higher the score, the heavier it is.We will decide whether to give psychological intervention based on the score.

CONTACTS AND LOCATIONS:
Locations (1):
- Feng, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No